CLINICAL TRIAL: NCT01351844
Title: Computer Based Educational Module for the Reduction of Arthralgia Syndrome Associated With Endocrine Therapy for Breast Cancer
Brief Title: The CEASE Study: Computer Based Educational Module for the Reduction of Arthralgia Syndrome Associated With Endocrine Therapy for Breast Cancer
Acronym: CEASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient patients
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Victoria Shanmugam, Associate Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-548
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer; Arthralgia
Keywords: Aromatase inhibitor; Arthralgia Syndrome; Exercise
MeSH Terms: conditions — Breast Neoplasms; Arthralgia; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and exercise intervention (Active Comparator): The "intervention" module will contain a brief series of slides with a voice-over. An occupational therapist will review recommended exercises.
  Interventions: Behavioral: Education and exercise intervention
- Education and general exercise (Placebo Comparator): The "control" module will contain a brief series of slides with a voice-over. A physical therapist with experience in treating breast cancer patients will demonstrate a series of 4-5 general stretching and toning exercises.
  Interventions: Behavioral: Education and General Exercise

INTERVENTIONS:
Behavioral: Education and exercise intervention — An occupational therapist who has clinical experience in hand therapy for breast cancer patients with arthralgia syndrome, will review 4-5 exercises which improve hand range of motion and reduce hand stiffness.
  Arms: Education and exercise intervention
Behavioral: Education and General Exercise — A physical therapist with experience in treating breast cancer patients with lymphedema will demonstrate a series of 4-5 general stretching and toning exercises.
  Arms: Education and general exercise

SUMMARY:
Patients have been asked to participate in the CEASE study because their treating oncologist has recommended that they start an aromatase inhibitor medication. These medications are associated with joint complaints. The purpose of this study is to see whether a computer-based educational module is a feasible intervention to help address these symptoms. If the patients agree to participate, a research coordinator will test their grip strength and give them a computer log-on code. They will be shown how to log-on to complete the educational module and a few simple questionnaires. Patients have the option to do this from home if they wish. In 3 months time, the investigators will ask patients to return to the clinic and have another grip strength evaluation and complete some additional questionnaires. The computer module and the follow up visit will each take about 30 minutes of time.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal stage I-III breast cancer patients
* Starting or about to start aromatase inhibitor
* English speaking with ability to read, write and use a computer to watch and listen to an educational module.
* Able to give informed consent

Exclusion Criteria:

* Aromatase inhibitor (AI) use for more than 6 months
* Metastatic breast cancer
* Non-English speaking, or unable to read, write or use a computer to watch and listen to an educational module.
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 3 months
  This study is designed as a pilot study to assess feasibility of this educational intervention in a small population of only 40 patients. Patients will be given the option to complete the module from home. The primary endpoint will be patient completion of the educational module and follow-up questionnaires.

SECONDARY OUTCOMES:
Grip Strength | 3 months
  The impact of the exercise education on symptoms will be assessed using grip strength evaluation with dynamometer at the baseline and three month follow-up visits, along with standardized pain and quality of life questionnaires completed at both time points.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria K Shanmugam, MD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Victoria Shanmugam, Washington D.C., District of Columbia, United States